CLINICAL TRIAL: NCT04675294
Title: A Phase 2 Study of ALX148 in Combination With Pembrolizumab in Patients With Advanced Head and Neck Squamous Cell Carcinoma (ASPEN-03)
Brief Title: Evorpacept (ALX148) in Combination With Pembrolizumab in Patients With Advanced Head and Neck Squamous Cell Carcinoma (ASPEN-03)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ALX Oncology Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT148003; KEYNOTE-B87 (Other: Merck Sharp & Dohme LLC); MK-3475-B87 (Other: Merck Sharp & Dohme LLC); 2020-004093-21 (EudraCT Number); 2023-508340-22-00 (EU CTIS Number)
Record Dates: First submitted 2020-12-15; First posted 2020-12-19 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma
Keywords: ALX148; CD47; SIRPα; HNSCC; pembrolizumab; evorpacept
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — ALX148; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- evorpacept (ALX148) + pembrolizumab (Experimental): evorpacept (ALX148) 45 mg/kg IV and pembrolizumab 200 mg IV given every 3 weeks.
  Interventions: Drug: evorpacept; Drug: pembrolizumab
- pembrolizumab (Active Comparator): pembrolizumab 200 mg IV given every 3 weeks.
  Interventions: Drug: pembrolizumab

INTERVENTIONS:
Drug: evorpacept — IV Q3W
  Other Names: ALX148
  Arms: evorpacept (ALX148) + pembrolizumab
Drug: pembrolizumab — IV Q3W
  Other Names: KEYTRUDA®

SUMMARY:
A Phase 2 Study of evorpacept (ALX148) in Combination With pembrolizumab in Patients With Advanced Head and Neck Squamous Cell Carcinoma.

DETAILED DESCRIPTION:
This is a open-label, randomized phase 2 multi-center study of the anti-tumor efficacy of evorpacept (ALX148) + pembrolizumab and of pembrolizumab alone in patients with metastatic or unresectable, recurrent HNSCC that is PD-L1 positive (CPS ≥1 by an FDA-approved test) and who have not yet been treated for their advanced disease. The study comprises an initial safety lead-in cohort followed by a randomized portion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic or unresectable, recurrent head and neck squamous cell carcinoma (HNSCC) that is PD-L1 positive (CPS > 1) and who have not received prior systemic therapy for their advanced disease.
* Adequate bone marrow function.
* Adequate renal and liver function.
* Adequate ECOG performance status.

Exclusion Criteria:

* Patients with known symptomatic CNS metastases or leptomeningeal disease requiring steroids.
* History of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Prior treatment with any anti-CD47 or anti-SIRPα agent.
* Prior treatment with anti-PD-1 or PD-L1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate per RECIST 1.1 | Last randomized patient reaching at least 24 weeks of follow-up

SECONDARY OUTCOMES:
Duration of response | Up to 36 months
Progression-free survival | Up to 36 months
Overall survival | Up to 36 months
Adverse events | Up to 36 months

CONTACTS AND LOCATIONS:
Locations (53):
- United States (14):
  - Hoag Hospital, Irvine, California
  - University of California San Diego, La Jolla, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Northwest Georgia Oncology Centers, Marietta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Blessing Cancer Center, Quincy, Illinois
  - University of Maryland Medical System, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Rutgers Cancer Institute of New Jersey, Newark, New Jersey
  - Memorial Sloan-Kettering Cancer Center, Long Island City, New York
  - The Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Vanderbilt - Ingram Cancer Center, Nashville, Tennessee
  - Houston Methodist Cancer Center, Houston, Texas
- Australia (5):
  - St. Vincent's, Sydney, New South Wales
  - Royal Brisbane and Womens Hospital, Brisbane, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Perth, Western Australia
  - Ashford Cancer Centre Research, Windsor Gardens
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
- Canada (4):
  - Hamilton Health Sciences - Juravinski Cancer Centre, Hamilton, Ontario
  - LHSC - Victoria Hospital, London, Ontario
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
- Netherlands (2):
  - VUMC Goederenontvangst, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
- Singapore (2):
  - National University Cancer Institute, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (14):
  - Chungbuk National University Hospital, Cheongju-si
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - CHA University of Bundang, Gyeonggi-do
  - Gachon University - Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Korea University Medical Center (KUMC) - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea - Eunpyeong St. Mary's Hospital, Seoul
  - Samsung Medical Center, Seoul
  - SNU Boramae Medical Center, Seoul
  - Severance Hospital Yonsei University, Seoul
  - Catholic University of Korea, St. Vincent's Hospital Suwon, Suwon
  - Yonsei University - Wonju Severance Christian Hospital, Wŏnju
- Spain (7):
  - Hospital Universitari Dexeus, Barcelona, Barcelona
  - Institud Catala d´Oncologia, Barcelona
  - Hospital Universitario La Paz, Madrid
  - HM Sanchinarro, Madrid
  - Hospital Severo Ochoa, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario de Navarra, Pamplona
- United Kingdom (2):
  - Royal Marsden NHS Foundation Trust, London
  - Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: No